CLINICAL TRIAL: NCT04036357
Title: Progression of LIver Damage and Cardiometabolic Disorders in Non-alcoholic Fatty Liver dIsease: an Observational Cohort STUDY. The Plinio Study
Brief Title: Liver Damage and Cardiometabolic Disorders in NAFLD
Acronym: PLINIO
Status: Recruiting | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Violi, Department Head, University of Roma La Sapienza
Other Study IDs: 2277/2011
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: NAFLD; Liver Fibroses; Cardiovascular Diseases; Cardiovascular Risk Factor
Keywords: NAFLD; Liver fibrosis; Cardiovascular
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Liver fibrosis is the most important prognostic factor in patients with non-alcoholic factor disease. Clinical and biological condition, as diabetes or mutation for PNPLA3, are well known factors associated with liver fibrosis onset and progression. However, little is known about biochemical factors predicting liver fibrosis evolution in large NAFLD populations.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is a common liver disease worldwide. NAFLD includes a spectrum of diseases raging from simple steatosis to non-alcoholic steatohepatitis (NASH), cirrhosis and hepatocellular carcinoma.

The prevalence of NAFLD ranges from 20% in the general population to 80-90% in obese and/or diabetic patients. Type 2 diabetes is also associated with disease progression. Some genetic conditions are known to be related with NAFLD pathophysiology. Mutation of patatin like phospholipase domain containing 3 (PNPLA3) is the most frequent genetic disorder associated with NAFLD onset and its accelerated progression. Both type 2 diabetes and PNPL3 mutation are the better-known factors associated with liver fibrosis.

More than the amount of lipid accumulation in the hepatocytes or of liver inflammation, the most important prognostic factors in NAFLD is fibrosis, which can occur in all stage of NAFLD disease, also in simple steatosis without inflammation or ballooning. Advanced fibrosis (F stage ≥ 3) has been related not only with liver-related death but also with death from all causes.

In 2007 a noninvasive system, the NAFLD fibrosis score (NFS), was validated to identify NAFLD patients with advanced fibrosis. NFS ≥ 0.676 detects an advanced fibrosis (F3-F4) with a positive predictive value of 90%-82% while NFS ≤ -1.455 excludes advanced fibrosis with a negative predictive value of 93%-88%.

In addition, in different settings, a score named Fibrosis-4 (FIB-4) was also validated to detect advanced fibrosis in patients with hepatitis B virus and hepatitis C virus /human immunodeficiency virus coinfection. Fib-4 ≤ 1.45 excludes advanced fibrosis with a negative predictive value of 90%, while Fib-4 ≥ 3.25 detects advanced fibrosis with a positive predictive value of 65%.

Currently, little is known about biochemical and pharmacological factors predicting liver fibrosis evolution in large cohorts of NAFLD patients.

Therefore, the primary aim of the study Is to investigate biochemical and pharmacological factors associated with fibrosis progression, identified as variations in noninvasive fibrosis scores, in a large population of patients with ultrasonography diagnosis of fatty liver disease.

A growing number of evidences show a higher cardiovascular risk in patients with NAFLD. Most of the data are derived from diabetic patients and there are not data derived from ad hoc studies. In addition, there are only few data on factors predicting incident cardiovascular (CV) events in patients with NAFLD.

Therefore, the secondary objective of the study is to investigate the association between NAFLD and CV events and to detect factors predicting CV events inception.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years old or more
* Patients with at least on of the following metabolic disorders

  * Obesity
  * Diabetes
  * Arterial hypertension
  * Dyslipidemia

Exclusion Criteria:

* Average daily consumption of alcohol >20 g in women and of >30 g in men (assessed by Alcohol Use Disorders Identification Test, AUDIT;
* presence of hepatitis B surface antigen and antibody to hepatitis C virus;
* positive tests for autoimmune hepatitis;
* cirrhosis and other chronic liver diseases;
* diagnosis of oncological diseases
* concomitant therapy with drugs known to promote liver steatosis (e.g. amiodarone);
* other chronic infectious or autoimmune disease;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive outpatients referring to the Day Service of Internal Medicine and Metabolic Diseases of the Department of Internal Medicine of Sapienza University of Rome for the management of cardio-metabolic risk factors, such as metabolic syndrome, dyslipidemia, hypertension, diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2011-11 (Actual); Primary Completion 2036-12-31 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical, biochemical and genetic factors associated to progression of liver fibrosis in a large cohort of patients with NAFLD | Patients will be followed for an expected mean time of 120 months
  To detect non conventional factors associated with the progression of liver fibrosis in patients with NAFLD. Progression of liver fibrosis will be assessed by non invasive markers (such as FIB-4, Nafld Fibrosis Score e liver elastography). The predictive role of the following factors will be assessed: plasmatic and urinary isoprostanes, thromboxane, platelet recruitment, reactive species of oxygen, nadph oxidase (nox2). Genes of interested will be sequenced.

SECONDARY OUTCOMES:
The predictive role of non-invasive markers of fibrosis on the incidence of major cardiovascular events. | Patients will be followed for an expected mean time of 60 months
  Non invasive score of liver fibrosis (such as NAFLD fibrosis score, AST-to-Platelets index and FIB-4) will be calculated at baseline and their predictive role on the incidence of major cardiovascular events will be tested
Nutritional factors associated to NAFLD | At Baseline
  Data on mediterranean diet adherence and on nutrients consumption will be collected and related to NAFLD severity. Data on circulating free fatty acid will be collected.
Platelet activation in NAFLD and NASH | At Baseline
  Plasmatic and urinary thromboxane and platelet recruitment will be measured as markers of platelets activation. Differences of these markers in different degree of NAFLD severity will be investigated
The predictive role of systemic markers of oxidative stress and antioxidant status on the incidence of cardiovascular events in NAFLD patients | Patients will be followed for an expected mean time of 120 months
  Oxidative stress markers such as plasmatic and urinary isoprostanes, thromboxane, platelet recruitment, reactive species of oxygen, nadph oxidase(nox2) will be measured. The predictive role of these markers on the incidence of cardiovascular events will be tested
Factors associated with chronic kidney disease in NAFLD patients | At Baseline
  To investigate the prevalence of chronic renal failure in Patients with NAFLD. Moreover, genetic, pharmacological and biochemical factors associated with estimated glomerular filtration rate (eGFR) < 90 and with eGFR < 60 will be investigated.
Predictors of kidney disease progression in patients with NAFLD | Patients will be followed for an expected mean time of 60 months
  The rate of Kidney disease progression in patients with NAFLD will be measured and will and compared to that in general populations. Predictors of kidney disease progression will be investigated.
Role of gut microbiota in NAFLD | At Baseline
  Serum Lipopolysaccharide (LPS) and serum zonulin will be measured in NAFLD patients and the correlation between LPS and NAFLD severity will be tested
Echocardiographic changes in patients with NAFLD | At Baseline
  Measures of systolic and diastolic function will be collected at baseline and correlated with the severity of NAFLD, of metabolic disorders and with genetic mutations correlated with NAFLD.
Score of cardiovascular risk in patients with NAFLD | Patients will be followed for an expected mean time of 120 months
  Performance of classical scores of cardiovascular risk will be tested in patients of NAFLD. In particular, the 2MACE score and the Systemic Coronary Risk Estimation (SCORE) will be tested. 2MACE score will be calculated assigning 2 points for Metabolic Syndrome and Age ≥75, 1 point for MI/revascularization, Congestive heart failure (ejection fraction ≤40 %), thrombo-Embolism (stroke/transient ischemic attack. The score, ranging from 0 to 7 points, will be considered positive for values higher than 2. SCORE will be calculated using age, sex, systolic blood pressure, smoking status, total and HDL cholesterol. The SCORE system estimates the 10-year cumulative risk of a first fatal atherosclerotic event. In absence of a good performance of pre-existing scores, we'll try to assess a specific cardiovascular risk score in NAFLD patients.
Dyslipidemia and cardiovascular events in patients with NAFLD | Patients will be followed for an expected mean time of 120 months
  The predictive role of triglycerides rich lipoproteins and cholesterol remnants will be evaluated.
Plasmatic and urinary isoprostanes | At Baseline
  Plasmatic and urinary isoprostanes will be measured as markers of systemic oxidative stress and of antioxidant status in NAFLD and NASH. Differences of these markers in different degree of NAFLD severity will be investigated
Reactive species of oxygen in NAFLD and NASH | At Baseline
  Reactive species of oxygen will be measured as markers of systemic oxidative stress and of antioxidant status in NAFLD and NASH. Differences of these markers in different degree of NAFLD severity will be investigated
Nadph oxidase (nox2) activation in NAFLD and NASH | At Baseline
  Nadph oxidase (nox2) activation will be estimated as markers of systemic oxidative stress and of antioxidant status in NAFLD and NASH. Differences of these markers in different degree of NAFLD severity will be investigated

CONTACTS AND LOCATIONS:
Overall Officials: Maria Del Ben, MD, Study Director — University of Roma La Sapienza; Daniele Pastori, MD, Principal Investigator — University of Roma La Sapienza; Francesco Baratta, MD, Principal Investigator — University of Roma La Sapienza; Francesco Angelico, MD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Day Service of Internal Medicine and Metabolic Disorders - Policlinico Umberto I - Sapienza University of Rome, Rome, Italy

REFERENCES:
- [Derived] Baratta F, Bartimoccia S, Pastori D, Cocomello N, Cammisotto V, Castellani V, Nocella C, Forte M, Picchio V, Carnevale R, Desideri G, Pignatelli P, Violi F. Neutrophil cathepsin G and risk of cardiovascular events in patients with diabetes mellitus. Cardiovasc Diabetol. 2025 Nov 26;24(1):448. doi: 10.1186/s12933-025-03005-y. PMID 41299502
- [Derived] Baratta F, D'Erasmo L, Di Costanzo A, Umbro I, Pastori D, Angelico F, Del Ben M. Metabolic Syndrome but Not Fatty Liver-Associated Genetic Variants Correlates with Glomerular Renal Function Decline in Patients with Non-Alcoholic Fatty Liver Disease. Biomedicines. 2022 Mar 19;10(3):720. doi: 10.3390/biomedicines10030720. PMID 35327522
- [Derived] Baratta F, Pastori D, Angelico F, Balla A, Paganini AM, Cocomello N, Ferro D, Violi F, Sanyal AJ, Del Ben M. Nonalcoholic Fatty Liver Disease and Fibrosis Associated With Increased Risk of Cardiovascular Events in a Prospective Study. Clin Gastroenterol Hepatol. 2020 Sep;18(10):2324-2331.e4. doi: 10.1016/j.cgh.2019.12.026. Epub 2019 Dec 27. PMID 31887443